CLINICAL TRIAL: NCT02260037
Title: A Double-blind, Randomised, Placebo-controlled Single Increasing Dose Tolerance Study in Healthy Male Volunteers After Intranasal Application of Epinastine Nasal (Dosage: 0.035 mg (0.025 % Solution) - 0.42 mg (0.3 % Solution))
Brief Title: Dose Tolerance Study in Healthy Male Volunteers After Intranasal Application of Epinastine Nasal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 262.261
Record Dates: First submitted 2014-10-07; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (2):
- Epinastine nasal (Experimental): single rising doses
  Interventions: Drug: Epinastine nasal
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Epinastine nasal
  Arms: Epinastine nasal
Drug: Placebo
  Arms: Placebo

SUMMARY:
Safety, tolerability and pharmacokinetics

ELIGIBILITY:
Inclusion Criteria:

* All participants in the study should be healthy, range from 21 to 50 years of age and be within ± 20 % of their normal weight (Broca -Index)
* Subsequently each subject will have his medical history taken and will receive a complete medical examination (incl. blood pressure and pulse rate measurements) as well as a 12-lead ECG. Haematological, hepatic and renal function tests will be carried out in the laboratory (Bioscientia Ingelheim, Germany). The subjects will fast for 12 hours before collection of specimens for all laboratory evaluations. The above mentioned examinations will be performed within 14 days before the first administration of the test substance
* In accordance with good clinical practice (GCP) and the local legislation all volunteers will have given their written informed consent prior to admission to the study

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastro-intestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study
* Use of any drugs which might influence the results of the trial (≤ one week prior to administration or during the trial)
* Participation in another trial with an investigational drug (≤ two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (≥ 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within the last week before the study)
* Any laboratory value outside the reference range of clinical relevance

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2001-08; Primary Completion 2001-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with clinically relevant findings in vital signs | up to 8 days after drug administration
  blood pressure, pulse rate
Number of patients with clinically relevant findings in 12-lead ECG | up to 8 days after drug administration
Number of patients with adverse events | up to 8 days after drug administration
Number of patients with clinically relevant findings in laboratory parameters | up to 8 days after drug administration
Changes in rhinoscopy assessment | up to 8 days after drug administration

SECONDARY OUTCOMES:
Maximum measured concentration in plasma (Cmax) | up to 48 hours after drug administration
Time from dosing to the maximum concentration in plasma (tmax) | up to 48 hours drug administration
Area under the concentration-time curve in plasma (AUC) | up to 48 hours after drug administration
Terminal rate constant of in plasma (λz) | up to 48 hours after drug administration
Apparent terminal half-life in plasma (t1/2) | up to 48 hours after drug administration
Total mean residence time in the body (MRTtot) | up to 48 hours after drug administration
Total clearance in plasma after extravascular administration (CL/F) | up to 48 hours after drug administration
Apparent volume of distribution during the terminal phase (Vz/F) | up to 48 hours after drug administration
Amount excreted into urine (Ae) | up to 48 hours after drug administration
Renal clearance (CLR) | up to 48 hours after drug administration
Assessment of dose-proportionality of epinastine nasal | up to 48 hours after drug administration
  based on AUC and Cmax